CLINICAL TRIAL: NCT00037258
Title: Dyslipidemia and Risk of Cardiovascular Disease in Diabetic Men and Women
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Frank Hu, Professor of Nutrition and Epidemiology, Brigham and Women's Hospital
Other Study IDs: 1156; R01HL065582 (NIH)
Record Dates: First submitted 2002-05-16; First posted 2002-05-17 (Estimated); Last update posted 2014-04-01 (Estimated); Status verified 2014-03

CONDITIONS: Cardiovascular Diseases; Diabetes Mellitus, Non-insulin Dependent; Heart Diseases; Atherosclerosis; Diabetes Mellitus
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus, Type 2; Heart Diseases; Atherosclerosis; Diabetes Mellitus

SUMMARY:
To determine the role of dyslipidemia, markers of endothelial dysfunction genetic susceptibility, and dietary fat intake on the development of cardiovascular disease (CVD) complications in Type II diabetes mellitus.

DETAILED DESCRIPTION:
BACKGROUND:

The cardiovascular disease complications of Type II diabetes mellitus are a major public health problem. The research is designed to provide new information about the relation of specific biomarkers, genes, and diet on risk of CVD complications in the high-risk Type II diabetes mellitus population.

DESIGN NARRATIVE:

The study assesses biochemical markers of dyslipidemia and endothelial dysfunction, and omega-3 fatty acids in relation to risk of CVD among men and women diagnosed with type 2 diabetes in two large ongoing cohort studies, the Nurses Health Study (NHS) and Health Professionals Follow-up Study (HPFS). By 1998, 12,600 confirmed type 2 diabetic cases had already accumulated in the two cohorts. By the year 2002, 5,507 blood samples prospectively collected from persons with previously or newly diagnosed type 2 diabetes will be available for analyses. Using this unparalleled resource, the investigators will evaluate (1) The relationship between plasma levels of cell adhesion molecules (i.e. sICAM-1, sVCAM-1, E-selectin), diabetic dyslipidemia, and risk of CVD among diabetics; (2) the association between Lp(a) concentrations and risk of CVD among diabetics, independent of high triglycerides and low HDL; (3) the association between long-term intakes of omega-3 fatty acids and CVD risk in diabetes. The main NHS and HPFS grants will provide follow-up and documentation of CVD in addition to covariate information. Overall, the large size of these cohorts, the prospective design, the high follow-up rates, and the availability of archived blood specimens provide a unique opportunity to study the relationship between diabetic dyslipidemia and risk of CVD in an extremely cost-efficient and timely manner. In addition, these two cohorts provide an unusual opportunity to compare lipid profiles and endothelial markers of CVD between diabetic men and women.

ELIGIBILITY:
No eligibility criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-09; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Hu — Harvard University School of Public Health

REFERENCES:
- [Background] Hu FB, Cho E, Rexrode KM, Albert CM, Manson JE. Fish and long-chain omega-3 fatty acid intake and risk of coronary heart disease and total mortality in diabetic women. Circulation. 2003 Apr 15;107(14):1852-7. doi: 10.1161/01.CIR.0000062644.42133.5F. Epub 2003 Mar 31. PMID 12668520
- [Background] Goldberger AL, Peng CK, Lipsitz LA. What is physiologic complexity and how does it change with aging and disease? Neurobiol Aging. 2002 Jan-Feb;23(1):23-6. doi: 10.1016/s0197-4580(01)00266-4. No abstract available. PMID 11755014
- [Background] Tanasescu M, Cho E, Manson JE, Hu FB. Dietary fat and cholesterol and the risk of cardiovascular disease among women with type 2 diabetes. Am J Clin Nutr. 2004 Jun;79(6):999-1005. doi: 10.1093/ajcn/79.6.999. PMID 15159229
- [Background] Shai I, Rimm EB, Schulze MB, Rifai N, Stampfer MJ, Hu FB. Moderate alcohol intake and markers of inflammation and endothelial dysfunction among diabetic men. Diabetologia. 2004 Oct;47(10):1760-7. doi: 10.1007/s00125-004-1526-0. Epub 2004 Oct 22. PMID 15502925
- [Background] Jiang R, Schulze MB, Li T, Rifai N, Stampfer MJ, Rimm EB, Hu FB. Non-HDL cholesterol and apolipoprotein B predict cardiovascular disease events among men with type 2 diabetes. Diabetes Care. 2004 Aug;27(8):1991-7. doi: 10.2337/diacare.27.8.1991. PMID 15277429
- [Background] Skinner HG, Michaud DS, Giovannucci EL, Rimm EB, Stampfer MJ, Willett WC, Colditz GA, Fuchs CS. A prospective study of folate intake and the risk of pancreatic cancer in men and women. Am J Epidemiol. 2004 Aug 1;160(3):248-58. doi: 10.1093/aje/kwh214. PMID 15257998
- [Background] Schulze MB, Rimm EB, Shai I, Rifai N, Hu FB. Relationship between adiponectin and glycemic control, blood lipids, and inflammatory markers in men with type 2 diabetes. Diabetes Care. 2004 Jul;27(7):1680-7. doi: 10.2337/diacare.27.7.1680. PMID 15220246
- [Background] Schulze MB, Rimm EB, Li T, Rifai N, Stampfer MJ, Hu FB. C-reactive protein and incident cardiovascular events among men with diabetes. Diabetes Care. 2004 Apr;27(4):889-94. doi: 10.2337/diacare.27.4.889. PMID 15047644
- [Background] Choi HK, Willett WC, Stampfer MJ, Rimm E, Hu FB. Dairy consumption and risk of type 2 diabetes mellitus in men: a prospective study. Arch Intern Med. 2005 May 9;165(9):997-1003. doi: 10.1001/archinte.165.9.997. PMID 15883237
- [Background] Qi L, Rimm E, Liu S, Rifai N, Hu FB. Dietary glycemic index, glycemic load, cereal fiber, and plasma adiponectin concentration in diabetic men. Diabetes Care. 2005 May;28(5):1022-8. doi: 10.2337/diacare.28.5.1022. PMID 15855561
- [Background] Wang Y, Rimm EB, Stampfer MJ, Willett WC, Hu FB. Comparison of abdominal adiposity and overall obesity in predicting risk of type 2 diabetes among men. Am J Clin Nutr. 2005 Mar;81(3):555-63. doi: 10.1093/ajcn/81.3.555. PMID 15755822
- [Background] Schulze MB, Shai I, Rimm EB, Li T, Rifai N, Hu FB. Adiponectin and future coronary heart disease events among men with type 2 diabetes. Diabetes. 2005 Feb;54(2):534-9. doi: 10.2337/diabetes.54.2.534. PMID 15677512